CLINICAL TRIAL: NCT00285987
Title: Quality of Life After an Ambulatory Reconstruction of the Cruciate Ligament
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has never started
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000/282
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Rupture of the Cruciate Ligament

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Reconstruction of the cruciate ligament

SUMMARY:
Study to compare the quality of life after reconstruction of the cruciate ligament in hospitalized versus day-clinic patient

ELIGIBILITY:
Inclusion Criteria:

* rupture of the cruciate ligament

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be